CLINICAL TRIAL: NCT03822819
Title: Investigation of the Optimal Cocktailed Probiotics for Decolonization of Vancomycin-resistant Enterococci in Human Gut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University (Other); Delta Electronics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N201805035
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Vancomycin-Resistant Enterococci; Probiotics
Keywords: vancomycin-resistant entercocci; probiotics; microbiome analysis pipeline; next generation sequencing; decolonization; virulence gene

STUDY DESIGN:
Intervention Model Description: The study is going to be carried out with two groups in which participants are either administered with probiotic cocktail capsules or placebo capsules
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic cocktail capsules uptake (Experimental): Participants take two capsules of probiotic cocktail everyday for 30 days in a double-blinded masking. Stool samples will be collected before and after capsule uptake and be analyzed for VRE number and microbiota change.
  Interventions: Dietary Supplement: probiotic cocktail capsules
- placebo capsules uptake (Placebo Comparator): Participants take two capsules of placebo everyday for 30 days in a double-blinded masking. Stool samples will be collected before and after capsule uptake and be analyzed for VRE number and microbiota change.
  Interventions: Dietary Supplement: placebo capsules

INTERVENTIONS:
Dietary Supplement: probiotic cocktail capsules — Daily uptake of probiotic cocktail for three weeks
  Arms: probiotic cocktail capsules uptake
Dietary Supplement: placebo capsules — Daily uptake of placebo capsule for three weeks
  Arms: placebo capsules uptake

SUMMARY:
Vancomycin-resistant enterococci (VRE) has been a serious public health issue as an opportunistic pathogen and reservoir of antibiotic resistant genes. To reduce VRE carriage in human gut, investigators aim to look for effective probiotic cocktail to compete with VRE in human gut microflora via the technique of microbiome analysis pipeline (MAP). The probiotic cocktail gave by MAP result will be tested in a clinical trial, in which 80 subjects with VRE carriage will be enrolled and allocated randomly into two groups. Subjects in first group will be administered with probiotic cocktail capsules, and placebo capsules will be given to the second group in a double-blind manner. Stool samples will be collected from subjects before and after three weeks of probiotic/probiotic capsule uptake, and analyzed for VRE number and gut microflora changes to evaluate the efficacy of probiotic cocktail.

DETAILED DESCRIPTION:
Enterococci are one of the commensal gut flora in humans and have become an important pathogenic bacterium of opportunistic infection. Enterococci can cause severe infection when the patients become immunocompromised and subsequent serious problem in medical therapy because last line antibiotics could be ineffective. The incidences of vancomycin-resistant enterococci (VRE) have been increasing all over the world in recent years. VRE have become a global threat in human health and medical care because of the possible spreading of antibiotic resistance genes. So far probiotic bacteria have played various important roles in regulation of gut functions and some positive impact on diabetes, liver function impairment, and psychiatric disorders. Recently a few probiotic studies indicated that VRE could possibly be decolonized from human gut. However, it remains controversial because of different probiotic strains, dosages, durations of administrations, and study designs in these reports. Therefore, further in vitro studies and clinical trials are warranted for validation of the hypothesis that VRE could be decolonized by probiotic bacteria from human gut.

In the preliminary study using Microbiome analysis pipeline to dissect the NGS (next generation sequencing) data from the co-cultures of two VRE strains (Enterococcus faecium, Enterococcus faecalis) and ten TFDA (Taiwan Food and Drug Administration)-approved probiotic bacteria, investigators have confirmed that the mixture of the ten probiotic bacteria significantly suppressed the bacterial amounts of VRE during the in vitro co-cultures. The results will provide a formula of optimal cocktailed probiotics in which a specific combination of the selected probiotic bacteria could exert a maximal effect on suppression of growth of VRE.

First, An in vitro co-culture of VRE and the optimal cocktailed probiotics selected by Microbiome analysis pipeline will be conducted for validation of the results from the preliminary study. Gastric acid-resistant capsules containing the probiotic cocktail validated with in vitro co-culture model, will then be prepared in dosage of 10^10 CFU (Colony Forming Unit).

Second, in the proposed clinical trial, participants of age between 20 and 90-year-old will be selected and admitted to Taipei Medical University Hospital with isolated vancomycin-resistance enterococci (VRE) from their stools after hospitalization. Exclusion criteria in this study are individuals: (1) with routine probiotic uptake in daily life, or being prescribed with probiotics in clinic one-week before or in the period of clinical trial; (2) being prescribed with oral antibiotic uptake in the period of clinical trial; (3) with diarrhea symptom; (4) in pregnancy; (5) of immuno-compromised conditions or being prescribed with steroid-type medicines; (6) with diabetes mellitus; (7) critically ill patients.

When the conditions of their underlying diseases are stabilized, these patients who sign the informed consents will be randomly assigned into two groups receiving the cocktailed probiotics or placebo for 3 weeks in double-blind masking. The stool samples will be collected before and after the 3-week administration of the cocktailed probiotics or placebo. After completion of enrolling 80 patients in total umber, the double-blinded capsules will be unlabeled and at least 50 patients with 25 completed paired stool samples in both groups will be further processed for genomic DNA isolation and 16s rDNA (ribosomal DNA) NGS analysis. Finally, the quantities of VRE in stool samples will be analyzed with colony formation number on selective medium, and alterations of gut microbiota will be analyzed through stool microbiome 16s rDNA NGS. The results will be compared between the cocktailed probiotics group and the placebo group for evaluation of the VRE decolonization effect of probiotics.

ELIGIBILITY:
Inclusion Criteria:

* VRE-carriage
* of age between 20 and 90-year-old
* agreeing to participate

Exclusion Criteria:

* routine probiotic uptake in daily life, or being prescribed with probiotics in clinic one- week before or in the period of clinical trial
* being prescribed with oral antibiotic uptake in the period of clinical trial
* with diarrhea symptom
* in pregnancy
* of immuno-compromised conditions or being prescribed with steroid-type medicines
* with diabetes mellitus
* critically ill patients

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
VRE number change | after 30 days of capsules uptake
  Stool samples will be collected from participants before and after capsule uptake and plating out on selective medium for VRE after proper serial dilution. VRE number is defined as VRE CFU per gram of stool sample, and compared between two samples from the same participant.

CONTACTS AND LOCATIONS:
Overall Officials: Shiuh-Bin Fang, M.D, Ph.D., Principal Investigator — Taipei Medical University-ShuangHo Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan